CLINICAL TRIAL: NCT03823872
Title: Effects of Eight Weeks of Concurrent Exercise Training and Time-restricted Feeding (16/8) on Body Composition, Muscle Endurance, Metabolism, Cardiovascular Risk Factors, and Dietary Intake in Males and Females.
Brief Title: Exercise Training and Time-restricted Feeding in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyle Hackney (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor-Investigator, Kyle Hackney, Assistant Professor, North Dakota State University
Organization: North Dakota State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE18247
Record Dates: First submitted 2018-11-10; First posted 2019-01-31 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Overweight and Obesity; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overweight (Experimental): Participants with BMI 25-29.9 kg/m2 undergo structured exercise for weight loss. They are randomized to the following interventions: 1) time restricted feeding = only eat between 12pm-8pm or 2) normal feeding= eat on normal schedule.
  Interventions: Other: Time restricted feeding; Other: Normal feeding
- Obese (Experimental): Participants with BMI 29.9-34.9 kg/m2 undergo structured exercise for weight loss. They are randomized to the following interventions: 1) time restricted feeding = only eat between 12pm-8pm or 2) normal feeding= eat on normal schedule.
  Interventions: Other: Time restricted feeding; Other: Normal feeding

INTERVENTIONS:
Other: Time restricted feeding — Time restricted feeding= consume food only from 12:00pm-8:00pm
Other: Normal feeding — Normal feeding= consume food per normal schedule

SUMMARY:
Overweight and obesity prevalence in adolescents and adults continues to remain significantly high in the United States. While diet and exercise improve many consequences of obesity, dietary strategies are not always nutrient sufficient and manageable long-term. Thus, highly complaint dietary strategies that lead to fat loss, while maintaining muscle mass, are needed. Time-restricted feeding (TRF) may be an ideal dietary approach for reducing fat mass and cardiovascular disease risk, while diminishing the loss of muscle mass and strength associated with obesity and aging. TRF, unlike continuous energy restriction, does not require a restrictive energy intake10. TRF requires individuals to consume calories within a set window of time (example = 8 hours), inducing a fasting window of 16 hours per day. There are few human studies on TRF that measure their effects in combination with both aerobic and resistance training. One recent study found an 8-hour TRF program (16-hour fast) improved insulin sensitivity, decreased fat mass, and maintained muscle mass in resistance-trained males after 8 weeks. Thus, the feasibility of TRF as dietary approach should be investigated further.The aims of this study are to: 1) determine whether time-restricted feeding (TRF) is an effective dietary strategy for reducing fat mass while preserving fat-free mass with aerobic and resistance training; 2) evaluate potential changes in health-related biomarkers (cardiovascular profile and anabolic-catabolic hormones) and muscle health indicators (mass, strength and quality) after 8 weeks of concurrent training with TRF; and 3) examine the influence of caloric intake and macronutrient consumption on muscle health in the TRF and normal feeding (NF) groups pre- to post-concurrent resistance training.

DETAILED DESCRIPTION:
Overweight and obesity prevalence in adolescents and adults continues to remain significantly high in the United States in all socioeconomic categories, regardless of racial and ethnic backgrounds. This is important because aging is strongly linked with increases in adiposity and alterations to the distribution of fat in the body, including visceral, hepatic, and intermuscular fat stores. These areas of fat storage are independently associated with increased risk of cardiovascular disease (CVD) and physical dysfunction. These conditions represent a major health problem in the US and are often triggered by multilayered dietary imbalances and lack of physical activity.

CVD is the leading cause of death in the United States, with 30% of adults older than 19 years of age having hypertension, and 16.5% of all deaths being attributed to high blood pressure. Physical disfunction with aging, also referred to as sarcopenia and dynapenia, is the gradual and progressive loss of muscle mass, strength, and endurance. Sarcopenia is characterized by a 3-8% loss of muscle mass per decade after the age of 30 years, affecting 30% of individuals over 60 years and 50% of individuals over 80 years. This age-related decline in muscle mass negatively affects strength, balance, and stability; leading to an increased risk of falls and impaired ability to perform activities of daily living such as walking, personal care, cooking, and chores. The most alarming consequence of decreased muscle strength is its ability to predict future mortality in middle-aged and older adults. While diet and exercise improve many health consequences of obesity and attenuate declines in muscle mass and strength, dietary strategies are not always nutrient sufficient and manageable for long-term use. Thus, highly compliant dietary strategies that facilitate fat loss while maintaining fat-free mass are needed.

Continuous energy restriction (CER), a reduction in daily caloric intake up to 40%, is a primary dietary strategy to help individuals decrease fat mass and lower the risk of CVD. While CER can be effective, it is associated with poor compliance and appears to accelerate the return of pre-deprivation body mass levels once the restraints over feeding are removed. More importantly, CER is known for weight loss consisting of up to 10%-60% fat-free mass, which suggests a large proportion of metabolically active skeletal muscle tissue is lost instead of adipose tissue. TRF, a variant of intermittent fasting, is an increasingly popular dietary approach because it does not require a restrictive energy intake as with CER. TRF allows individuals to consume ad libitum energy intake within a set window of time (example = 8 hours), inducing a fasting window of 16 hours per day. Literature from animal studies have demonstrated reductions in body weight, total cholesterol, and concentrations of triglycerides, glucose, insulin, as well as improvements in insulin sensitivity following TRF. Unfortunately, human studies on TRF are limited and few exist that measure their effects in combination with aerobic or resistance training.

One recent study recruited 34 healthy, resistance-trained males and randomized them into either a TRF (16-hour fast) or NF group. The groups were tested before and after eight weeks of their diet assignment and standardized resistance training for body composition, maximal strength, and multiple health-related biomarkers. These biomarkers included total and free testosterone, IGF-1, blood glucose, insulin, adiponectin, leptin, triiodothyronine (T3), thyroid stimulating hormone, interleukin-6, interleukin-1B (IL-1B), tumor necrosis factor a (TNF-a), total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides. After the eight weeks of training, the TRF group significantly decreased fat mass compared to a NF group (-16.4% vs -2.8%). Hormonal responses included significantly reduced levels of total testosterone and IGF-1 with TRF, typically seen during CER. Though these anabolic hormones were reduced, no reductions in fat-free mass and strength were observed. In fact, fat-free mass, as well as arm and thigh cross-sectional area, was maintained in both groups. Leg press one-repetition maximum increased significantly in both groups, and, while not significant, bench press one-repetition maximum increased in both groups. These increase in strength are important to note, considering the subjects were highly resistance trained. Another interesting effect of TRF was reduced blood glucose and insulin levels, which contributed to a significant improvement in HOMA-IR (insulin resistance). Adiponectin increased, while leptin decreased with TRF. These responses were said to be linked to an enhanced regulation of insulin sensitivity and an improved anti-inflammatory effect in the TRF group. Lastly, T3 and Triglycerides decreased significantly and TNF-a and IL-1B were lower in TRF compared to NF. Overall, the study established TRF as a beneficial dietary strategy to improve health-related biomarkers, decrease fat mass, and maintain fat-free mass. Therefore, the feasibility of TRF as a dietary approach, for improving body composition and attenuating the risk factors of CVD and physical dysfunction that occur with obesity and aging, should be investigated further.The study will recruit 40, overweight (determined by body mass index between 25.0-29.9 kg/m2) male and female participants (ages of 45-60 years old) who are not currently following a structured aerobic or resistance training program or dietary plan. This will be a randomized, controlled trial with assessments made pre- and post-intervention. All subjects will be scheduled for an 8-week, standardized aerobic and resistance training program. Participants in TRF group will be required to consume all their energy intake in an 8-hour feeding window (12:00pm to 8:00pm), and will perform their exercise training within that feeding window. Participants in the NF group will maintain their typical dietary habits. Once training is finished, participants will complete post-training assessments that include all pre-training assessment variables.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index 25.0-34.9 kg/m2, generally healthy and mobile.

Exclusion Criteria:

* Currently smoke tobacco.
* e-cigarettes, or used smokeless tobacco.
* Diagnosed neuromuscular disease.
* Diagnosed diabetes,
* Diagnosed high blood pressure.
* Diagnosed cancer.
* Previous heart attack or other chronic heart related conditions.
* Difficulty moving without assistive devices.
* Difficulty walking one quarter mile.
* Taking medications that influence muscle size.
* Previous bariatric surgery.
* Greater than 350 lbs in body mass.
* Currently on a dietary or exercise program.
* At risk for disordered eating via self-report.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Body mass after 8 weeks | change from 8 weeks
  mass kg of subject on a calibrated scale
Change from Baseline fat mass after 8 weeks | change from 8 weeks
  fat mass in kg of the subject measured by DXA
Change from Baseline lean mass after 8 weeks | change from 8 weeks
  lean mass kg of the subject measured by DXA

SECONDARY OUTCOMES:
Change from Baseline insulin after 8 weeks | change from 8 weeks
  insulin µIU/mLvia blood spot testing
Change from Baseline high-sensitivity C-reactive protein (Hs-CRP) after 8 weeks | change from 8 weeks
  Hs-CRP in mg/Lvia blood spot testing
Change from Baseline hemoglobin A1c after 8 weeks | change from 8 weeks
  hemoglobin A1c % via blood spot testing
Change from Baseline triglycerides after 8 weeks | change from 8 weeks
  triglycerides in mg/dL via blood spot testing
Change from Baseline cholesterol 8 weeks | change from 8 weeks
  cholesterol mg/dL via blood spot testing
Change from Baseline HDL after 8 weeks | change from 8 weeks
  HDL mg/dL from blood spot testing
Change from Baseline LDL after 8 weeks | change from 8 weeks
  LDL mg/dL via blood spot testing
Change from Baseline VLDL after 8 weeks | change from 8 weeks
  VLDL mg/dL from blood spot testing
Change from Baseline estradiol after 8 weeks | change from 8 weeks
  estradiol pg/mL from saliva testing
Change from Baseline progesterone after 8 weeks | change from 8 weeks
  progesterone pg/mL from saliva testing
Change from Baseline testosterone after 8 weeks | change from 8 weeks
  testosterone pg/mL from saliva testing
Change from Baseline cortisol after 8 weeks | change from 8 weeks
  cortisol pg/mL from saliva testing
Change from Baseline lower body strength after 8 weeks | change from 8 weeks
  biodex assessment in Newtons
Change from Baseline upper body strength after 8 weeks | change from 8 weeks
  handgrip assessment in kg

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States